CLINICAL TRIAL: NCT01694446
Title: Regulation of Intestinal and Hepatic Lipoprotein Production by Glucose and Fructose
Acronym: glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Glucose 090428B
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hyperlipidemia
Keywords: Intestinal lipoprotein; Apo B48 and apoB100; Pancreatic clamp
MeSH Terms: conditions — Hyperlipidemias | interventions — Fructose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraduodenal glucose or fructose (Experimental)
  Interventions: Other: Intraduodenal glucose or fructose

INTERVENTIONS:
Other: Intraduodenal glucose or fructose

SUMMARY:
Increased postprandial plasma triglycerides are associated with increased cardiovascular risk. Chronic consumption of carbohydrates is associated with increased levels of triglycerides. Very few studies have assessed the effect of acute consumption of carbohydrates on plasma triglycerides and lipoprotein production and clearance. The present study aims to assess the effects of acute administration of glucose and fructose on hepatic and intestinal lipoprotein production.

DETAILED DESCRIPTION:
Each subject will be studied twice 4-6 weeks apart in random order in this single blinded study. A nasoduodenal tube will be sited under fluoroscopic guidance the day prior to the study.In study A they will receive intraduodenal intralipid (20% at 60 ml/hour) alongside 60 ml/hour of 20% dextrose or fructose for 15 hours starting at 4am. In study B they will receive 60 ml/hour of intraduodenal intralipid with 60ml/hour of normal saline for 15 hours from 4am. A pancreatic clamp (octreotide with replacement glucose, insulin, glucagon and growth hormone) will be started at 7am. From 9am an iv bolus of deuterated-glycerol (d5-glycerol) along with a regular infusion of deuterated leucine (L-[5,5,5-2H3]. Regular blood samples will be drawn to assess lipoprotein kinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20 kg/m2 to 27 kg/m2
3. Hemoglobin above 130g/L.
4. Normal glucose tolerance in response to a 75g, 2-hr OGTT

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. History of diabetes or OGTT indicative of diabetes or impaired glucose tolerance.
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
6. Current addiction to alcohol or substances of abuse as determined by the investigator.
7. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
8. Taking any prescription or non-prescription medications at the time of the study
9. Having donated blood three months prior to and three months post study procedures
10. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects. Those who test positive for pregnancy will be excluded.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assessment of intestinal and hepatic lipoprotein production | 10 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hopital, Toronto, Ontario, Canada